CLINICAL TRIAL: NCT01457781
Title: A Phase 2, Placebo Controlled, Double-Blind, Randomized, Clinical Study to Determine Safety, Tolerability and Efficacy of Pulsed, Inhaled Nitric Oxide (iNO) Versus Placebo as Add-On Therapy in Symptomatic Subjects With Pulmonary Arterial Hypertension (PAH)
Brief Title: Inhaled Nitric Oxide/INOpulse DS for Pulmonary Arterial Hypertension (PAH)
Acronym: PAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bellerophon Pulse Technologies (Industry)
Responsible Party: Sponsor
Organization: Bellerophon (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IK-7001-PAH-201
Record Dates: First submitted 2011-10-12; First posted 2011-10-24 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Hypertension
Keywords: Inhaled nitric oxide; pulmonary arterial hypertension; pulmonary hypertension; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.025 mg inhaled nitric oxide (Active Comparator): Inhaled nitric oxide (iNO) 0.025 mg/kg IBW/hr for up to 24 hours/day x 16 weeks (3.0 mg/L [2440 ppm] NO mini-cylinder; change q 24 hours) delivered via INOpulse® DS delivery device.
  Interventions: Combination Product: Inhaled Nitric Oxide 0.025 mg/kg IBW/hr delivered via INOpulse DS Device
- 0.075 mg inhaled nitric oxide (Active Comparator): Inhaled nitric oxide (iNO) 0.075 mg/kg IBW/hr for up to 24 hours/day x 16 weeks (6.0 mg/L [4880 ppm] NO mini-cylinder; change q 24 hours) delivered via INOpulse® DS delivery device.
  Interventions: Combination Product: Inhaled nitric oxide 0.075 mg/kg IBW/hr delivered via INOpulse DS Device
- placebo (Placebo Comparator): Placebo 0.075 mg/kg IBW/hr for up to 24 hours/day x 16 weeks* (99.999% Nitrogen [N2] mini-cylinder; change q 24 hours) delivered via INOpulse® DS delivery device.
  Interventions: Combination Product: Placebo delivered via INOpulse DS Device

INTERVENTIONS:
Combination Product: Inhaled Nitric Oxide 0.025 mg/kg IBW/hr delivered via INOpulse DS Device — Cohort 1: 0.025 mg/kg IBW/hr for up to 24 hours/day x 16 weeks (3.0 mg/L [2440 ppm] NO mini-cylinder; change q 24 hours) delivered via INOpulse DS Device and INOpulse DS nasal cannula
  Arms: 0.025 mg inhaled nitric oxide
Combination Product: Placebo delivered via INOpulse DS Device — Placebo 0.075 mg/kg IBW/hr for up to 24 hours/day x 16 weeks (Nitrogen N2, 99.999%) delivered via INOpulse DS Device and INOpulse DS nasal cannula
  Arms: placebo
Combination Product: Inhaled nitric oxide 0.075 mg/kg IBW/hr delivered via INOpulse DS Device — Cohort 2: 0.075 mg/kg IBW/hr for up to 24 hours/day x 16 weeks (6.0 mg/L [4880 ppm] NO mini-cylinder; change q 24 hours) delivered via INOpulse DS Device and INOpulse DS nasal cannula
  Arms: 0.075 mg inhaled nitric oxide

SUMMARY:
This is a Phase 2, Placebo Controlled, Double-Blind, Randomized, Clinical Study to Determine Safety, Tolerability and Efficacy of Pulsed, Inhaled Nitric Oxide (iNO) Versus Placebo as Add-on Therapy in Symptomatic Subjects with Pulmonary Arterial Hypertension (PAH).

DETAILED DESCRIPTION:
Study to determine if inhaled nitric oxide (iNO) given through a special delivery device (INOpulse® DS) is safe and efficacious in treating Pulmonary Arterial Hypertension (PAH). Medical literature and clinical experience suggests that iNO at pulsed doses of 0.013 to 0.1 mg/kg per hour for 1 month to 2+ years appears safe and suggests efficacy for the treatment of pulmonary hypertension.

There are two parts to this study. In Part 1 (week 0 to week 16), the objectives are to determine the safety, tolerability, efficacy, and exploratory objectives of two different doses of iNO delivered by a pulsed delivery device in symptomatic subjects with PAH who remain symptomatic due to PAH on approved PAH monotherapy or combination approved PAH therapy. In Part 2 (week 17 to end of study Part 2 [EOS Part 2]), the objective is to compile data on the long-term effects of iNO on safety, tolerability, clinical and hemodynamic measures.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF) (and assent as appropriate) prior to the initiation of any study mandated procedures or assessments
2. A confirmed diagnosis of Pulmonary Hypertension Group 1 (PAH) who have either idiopathic PAH (IPAH), heritable PAH, anorexigen-induced PAH, associated PAH (APAH) with connective tissue disease (CTD), APAH with repaired simple congenital systemic to pulmonary shunt (i.e., atrial septal defect [ASD], ventricular septal defect [VSD] and/or patent ductus arteriosus [PDA]; complete repair at least 1 year prior to Screening) or APAH with human immunodeficiency virus (HIV)
3. Confirmation of PAH diagnosis at the time of Baseline RHC according to the following definition: mPAP ≥ 25 mmHg at rest, with a concomitant mean pulmonary capillary wedge pressure (mPCWP), mean left atrial pressure (mLAP), or left ventricular end diastolic pressure (LVEDP) ≤ 15 mmHg and a PVR ≥ 240 dynes.sec/cm-5
4. 6MWD at least 100 meters and no greater than 450 meters
5. The subject is receiving at least one approved PAH therapy and is clinically symptomatic from PAH (e.g., onset or increased dyspnea on exertion, dizziness, near-syncope, syncope, chest pain or peripheral edema)
6. Background PAH medication doses (including calcium channel blockade if being used to treat PAH) must be stable for at least 12 weeks prior to Screening
7. If on background conventional therapy (e.g., digoxin, diuretics, supplemental oxygen, anticoagulation), it must have been started at least 30 days prior to Screening and be on a stable dose for at least 30 days except for anticoagulation dose
8. If previously treated with an endothelin receptor antagonist (ERA), phosphodiesterase-5 (PDE-5) inhibitor, prostacyclin or a prostacyclin analog and is no longer on said treatment at Screening (per inclusion criteria as above), subject must have been off said treatment for > 90 days at Screening
9. If previously treated with a calcium channel blocker as treatment for PAH and is no longer on the calcium channel blocker treatment at Screening (per inclusion criteria as above), subject must have been off the calcium channel blocker treatment for > 90 days at Screening
10. Age between 16 and 80 years (inclusive)
11. Male height ≤ 200 cm (6'7") or Female height ≤ 210 cm (6'11")
12. Subjects are willing and considered in the judgment of the Investigator able to use the INOpulse DS device continuously for up to 24 hours per day
13. Females of childbearing potential must have a negative pre-treatment serum pregnancy test and must be on a reliable method of contraception (including double protection if appropriate, e.g., for subjects concurrently treated with bosentan therapy)

Exclusion Criteria:

1. Subjects with known HIV infection within the past 2 years who have a history of or show any clinical or laboratory evidence of any opportunistic pulmonary disease (e.g., tuberculosis, Pneumocystis carinii pneumonia, or other pneumonias) at the time of Screening
2. PAH associated with portal hypertension, untreated thyroid disorders, glycogen storage disease, Gaucher's disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders or splenectomy
3. Any subject with unrepaired congenital heart disease or repaired congenital heart disease other than the simple congenital to systemic shunts specified in the inclusion criteria, i.e., PAH associated with non-corrected simple congenital systemic-to-pulmonary shunts, corrected simple congenital systemic-to-pulmonary shunt with residual shunt post repair, or complex systemic-to- pulmonary shunts, corrected or non-corrected, or any other complex congenital heart disease, corrected or non-corrected
4. PAH associated with significant venous or capillary involvement (PCWP > 15 mmHg), known pulmonary veno-occlusive disease, or pulmonary capillary hemangiomatosis
5. Any subject with WHO PH Groups 2, 3, 4 or 5
6. Left ventricular systolic dysfunction, i.e., left ventricular ejection fraction (LVEF) < 40% or left ventricular shortening fraction (LVSF) < 22%
7. Left ventricular diastolic dysfunction, i.e., PCWP > 15 mmHg at rest or with exercise, acute volume loading or pharmacologic testing
8. History of clinically significant cardiomyopathy or valvular heart disease (i.e., moderate or greater aortic insufficiency; moderate or greater aortic stenosis; or moderate or greater mitral valve disease)
9. Clinically significant cardiac ischemic disease requiring use of nitrates, or hospital admission for acute coronary syndrome or intervention (percutaneous coronary intervention, coronary artery stent, coronary artery bypass surgery) within the past 90 days
10. Down syndrome
11. Any subject who develops a PCWP > 20 mmHg during AVT with iNO
12. Systemic hypertension defined as systolic blood pressure (SBP) > 160 mmHg and/or diastolic blood pressure (DBP) > 100 mmHg persistent at Screening after a period of rest (treated or untreated)
13. Systemic hypotension defined as SBP < 90 mmHg persistent at Screening after a period of rest
14. Moderate to severe obstructive lung disease defined as both a forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) < 70% and FEV1 < 65% of predicted value (bronchodilator administration prior to testing is optional; the test should be done within 3 years for all subjects with the exception of APAH/CTD which needs to be done within 6 months prior to Screening)
15. Moderate to severe restrictive lung disease: total lung capacity (TLC) < 60% of predicted; if TLC 60% to 70% predicted, a high resolution CT scan showing diffuse disease or more than mild patchy disease (done within 3 years for all subjects with the exception of APAH/CTD which needs to be done within 6 months prior to Screening)
16. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C
17. Estimated creatinine clearance < 30 mL/min (Cockcroft-Gault formula)
18. Hemoglobin < 10 gm/dL at Screening or Baseline
19. Acute or chronic physical impairment (other than dyspnea due to PAH) that would limit the ability to comply with study procedures or adherence to therapy, including carrying and wearing the INOpulse device per study protocol
20. Pregnant or breast-feeding at Screening
21. Administered L-arginine within 30 days prior to Screening
22. Known concomitant life-threatening disease with a life expectancy less than 1 year
23. Recently started (< 12 weeks prior to randomization) or planned cardiopulmonary rehabilitation program to start within the 16 week controlled study
24. Atrial septostomy within 3 months of randomization
25. Any subject with PAH who is treatment naïve or receiving any unapproved therapy as their only PAH treatment (including calcium channel blockade if the calcium channel blockade is the only treatment for the PAH)
26. Any subject who requires the use of a continuous positive airway pressure (CPAP), bilevel positive airway pressure (BiPAP), or other positive pressure devices to treat obstructive sleep apnea
27. Medical problem(s) likely to preclude completion of Part 1
28. Use of investigational drugs or devices within 30 days prior to enrollment into the study (other than acute vasodilator testing with iNO or IV epoprostenol)
29. Any underlying medical or psychiatric condition that, in the opinion of the Investigator, makes the subject an unsuitable candidate for the study
30. Any condition other than the subject's PAH that, in that opinion of the investigator, affects their ability to perform the 6MWT
31. Refusal to follow the protocol, including the two RHCs in Part 1 and one RHC in Part 2
32. Unable to travel to the investigational site for all required study visits and for all additional visits per the judgment of the Investigator or Sponsor

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is change in pulmonary vascular resistance (PVR) (dynes. sec/cm-5) from baseline to EOS Part 1. | baseline to Week 16
  Change from Baseline to 18 weeks in PVR

SECONDARY OUTCOMES:
Change in 6 minute walk distance (6MWD) from baseline to EOS Part 1 | baseline to Week 16
  6MWT Change from Baseline to Week 16
Time (in days) to first clinical worsening event (TTCW) from randomization to EOS Part 1 | randomization to Week 16
  Time (in days) to first clinical worsening event (TTCW) from randomization to EOS Part 1
Change in World Health Organization (WHO) Functional Class from baseline to EOS Part 1 | baseline to Week 16
  WHO Functional Class Change from Baseline to Week 16
Change in Borg Dyspnea Score (BDS) from baseline to EOS Part 1 | baseline to Week 16
  BDS change in Baseline to Week 16
Change in patient reported outcome (PRO) scores by the SF-36 short form version 2 and the Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) from baseline to EOS Part 1 | baseline to Week 16
  Patient Reported Outcome change from Baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, MD, Study Director — Bellerophon Therapeutics
Locations (51):
- United States (47):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - Allianz Research Institute, Inc., Fountain Valley, California
  - University of California, San Francisco-Fresno, Fresno, California
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Med Ctr, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - South Denver Cardiology Associates P.C., Littleton, Colorado
  - Christiana Care Health System, Newark, Delaware
  - University of Florida College of Medicine, Jacksonville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University Hospital-Emory Clinic, Atlanta, Georgia
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Gill Heart, Lexington, Kentucky
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - LSUHSC-New Orleans, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University Medical Center/Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Cardiovascular Division, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Medicine and Dentistry of NJ, Newark, New Jersey
  - Barnabas Health Newark Beth Israel Medical Center, Newark, New Jersey
  - Beth Israel Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - UC Health/University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Martha Morehouse Medical Pavillion, Columbus, Ohio
  - South Oklahoma Heart Research LLC, Oklahoma City, Oklahoma
  - Legacy Medical Group - Pulmonary Clinic, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute/Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Sioux Falls Cardiovascular PC, Sioux Falls, South Dakota
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (4):
  - Peter Lougheed Center, Calgary, Alberta
  - ABACUS - University of Alberta Hospitals, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No